CLINICAL TRIAL: NCT05802524
Title: Neurophysiological Approach for the Evaluation of Residual Cognitive Functions in Patients With Severe Alterations of Consciousness
Brief Title: Neurophysiological Evaluation of Residual Cognitive Functions in Patients With Severe Alterations of Consciousness
Status: Completed | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Other Study IDs: Multi-NW
Record Dates: First submitted 2023-03-15; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Consciousness Disorder; Cognitive Impairment
MeSH Terms: conditions — Consciousness Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neurowave Group — Neurosensory stimulation will consist in the administration of pairs of stimuli consisting of emotionally significant images and sounds in the personal life history (two rare stimuli) alternating with neutral images and sounds devoid of emotional significance (two "distracting" stimuli

SUMMARY:
Identify potential markers of recovery through event-related potentials (ERPs) in the evolution of altered consciousness with potential ability to discriminate between different conditions of altered state of consciousness.

Identify potential markers with prognostic value, in order to identify personalized and specific intensive rehabilitation paths based on the outcome indexes obtained.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale (GCS) > 8;

Level of Cognitive Scale (LCF) = 1-3;

Signature of the consent from the family member and/or guardian.

Exclusion Criteria:

* Failure to sign the consent of the family member and/or legal guardian;

Patients with cranial anatomical alterations that do not allow the correct assembly of the electrodes, caps, etc.;

Patients with absence of neurophysiological responses in visual evoked potentials (VEP) and with absence of peripheral waves (I-II wave) to acoustic potentials (PEA).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Departments of Serious Acquired Brain Injuries
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Event-related evoked potentials(ERPs) | 24 months
  Event-related evoked potentials(ERPs) are variations of the electric potential deriving from a visual, somesthetic or auditory stimulus.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided
corresponding author